CLINICAL TRIAL: NCT03450135
Title: Ovarian Hormone Variability and Mood Symptoms in Girls During the Pubertal Transition
Brief Title: Neurophysiology, Estrogen, and Stress Exposure in the Emergence of Depression in Adolescent Girls
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2173; 2KR961702 (Other Grant/Funding Number: NIH Clinical and Translational Science Award (CTSA))
Record Dates: First submitted 2018-02-14; First posted 2018-03-01 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Adolescent Development; Stress; Emotional Disturbances
Keywords: puberty; EEG; estradiol; mood; stress
MeSH Terms: conditions — Affective Symptoms | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum samples will be stored to potentially assess neurosteroids and additional stress-responsive biomarkers in the future. Samples will be labelled by subject ID, without personal identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mid-pubertal girls: Adolescent girls (ages 11-14) who are undergoing a healthy pubertal transition (Tanner developmental stage 3 or 4) will perform Trier Social Stress Test and Emotional go/no-go task.
  Interventions: Behavioral: Trier Social Stress Test; Behavioral: Emotional go/no-go task

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Participants will perform an acute psychosocial stress manipulation (Trier Social Stress Test) involving a speech task and challenging mental arithmetic.
Behavioral: Emotional go/no-go task — Participants will perform an emotional go/no-go paradigm to examine electrophysiological (EEG) correlates of cognitive and affective processing.

SUMMARY:
The prevalence of adolescent depression is steadily rising in the U.S., especially among adolescent girls. Currently 20% of adolescent girls experience major depression compared with 6% of boys (National Institute of Mental Health, 2016). The profound gender disparity in depression that emerges at puberty, but not before, implicates a role of ovarian steroid hormones in promoting affective (mood) symptoms in adolescent girls. In addition to dramatic physical maturation and a rapidly changing reproductive hormone environment at puberty, adolescence is also a time of exposure to substantial psychosocial stress, particularly in girls. It is well documented that stress interferes with the maturation of neurodevelopmental trajectories and is a critical precipitating factor in the pathway to psychopathology. However, the neuropathophysiological mechanisms linking stress exposure and sensitivity to ovarian hormone fluctuations at puberty to the onset and maintenance of depression symptoms in adolescence have yet to be elucidated, and is the purpose of this research.

DETAILED DESCRIPTION:
Framed within a diathesis-stress model of disease, the primary objective of this research is to determine a pathophysiological role of estradiol (E2) variability in the context of severe psychosocial stress exposure in regulating neurophysiological correlates of affective state change in girls (ages 11-14) during the pubertal transition (i.e., Tanner developmental stages 3 or 4). The rationale for examining E2 variability as a diathesis for mood impairment is twofold. First, sensitivity to hormonal flux during specific reproductive events has been shown to trigger affective symptoms in susceptible women, and second, E2 is a powerful neuroregulator of neural networks implicated in depression.

55 peripubertal girls undergoing a healthy pubertal transition will be recruited for the study. Over an 8-week period, depression symptoms (Center for Epidemiological Studies Depression Scale for Children (CES-DC)), anxiety (State Trait Anxiety Inventory (STAI-C)), and perceived stress (perceived stress scale (PSS)), and salivary E2 measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS) will be assessed on a weekly basis. An electroencephalogram (EEG) during an emotional go/no-go task will be performed after the 8-week collection period to probe neurophysiological correlates of maturing fronto-limbic circuitry and assess key domains of cognitive and emotional processing impacted by the hormonal milieu. At the follow-up visit, an acute psychosocial stressor (Trier Social Stress Test) will be administered to examine cortisol and autonomic stress reactivity. The central hypothesis of the proposed research is that the amplitude and synchrony of frontal neural oscillations evoked during the cognitive-affective processing paradigm, and cortisol reactivity to the psychosocial stressor will partially mediate the relationship between greater E2 variability and elevated depression symptoms in peripubertal girls, and this relationship will be particularly strong in girls who have experienced recent (within six months) psychosocial stress.

ELIGIBILITY:
Inclusion Criteria:

* Female, 11 to 14 years of age
* Meet Tanner developmental stage criteria (as indicated by self-report and pictorial scales of breast and pubic hair development) for pubertal stages 3 or 4
* Must be undergoing a healthy pubertal transition, pre-or-post menarche (within 15 months of menarche, with cycle irregularity)
* Girls must be able to read at a 4th-grade reading level

Exclusion Criteria:

* Current suicidal intent (based off Columbia-Suicide Severity rating scale)
* A history or current diagnosis of bipolar disorder or psychosis
* Currently on any prescription medications

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study will recruit participants of various racial, ethnic and socioeconomic backgrounds, reflective of the local population (60% White, 20% Black or African American, 10% Asian, and 10% Hispanic or Latino). Participants will be recruited from medical offices, schools and community centers (youth groups, church groups) in Orange and Durham Counties.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Average mood symptom score from Mood and Feelings Questionnaire | Week 10
  The MFQ consists of 33 descriptive phrases regarding how the subject has been feeling or acting recently (past two weeks) on a 3-point force-choice Likert-type response scales (most of the time, sometimes, or not at all). Greater scores reflect greater symptom severity.

SECONDARY OUTCOMES:
Theta (4-8 Hz) oscillatory activity elicited during an affective task | Week 10
  Theta oscillations (synchronization of power and phase with respect to stimulus presentation) will be assessed during an emotional go/no-go paradigm to reflect cognitive and emotional processing.
Salivary cortisol response to an acute psychosocial stress manipulation | Week 10
  The stress hormone cortisol will be assessed at rest and in response to the Trier Social Stress Test at baseline (enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Andersen, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, SHARRP Lab, Chapel Hill, North Carolina, United States